CLINICAL TRIAL: NCT06140901
Title: Morphological and Functional Pilot Study of the Bronchial Epithelium of Children With Post-infectious Bronchiolitis Obliterans
Brief Title: Bronchial Epithelium of Children With Post-infectious Bronchiolitis Obliterans
Acronym: e-PIBO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C23-37; 2023-A01544-41 (Other: IDRCB Number)
Record Dates: First submitted 2023-10-27; First posted 2023-11-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Bronchiolitis Obliterans
Keywords: children; post infectious
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective longitudinal study (AP-HM), in children aged 1 month to 6 years, comparing children hospitalized for lower respiratory infection by ADV or RV progressing or not to PIBO.
  After inclusion of the patients, a second nasal swab will be taken as part of the research for the PCR study of the subtypes of the virus responsible for the viral infection. Following the diagnosis of PIBO, bronchial endoscopy for microbiology and bronchial biopsies will be performed as part of routine care to rule out differential diagnoses. During this endoscopy, 2 additional bronchial biopsies and nasal brushing for research will be performed to recover epithelial cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm non PIBO (Active Comparator): children hospitalized for adenovirus or rhinovirus infection with non progressing to PIBO
  Interventions: Diagnostic Test: Study morphological and functional of respiratory epithelium
- Arm PIBO (Active Comparator): Children hospitalized for adenovirus or rhinovirus infection with progressing to PIBO in evolution.
  Interventions: Diagnostic Test: Study morphological and functional of respiratory epithelium

INTERVENTIONS:
Diagnostic Test: Study morphological and functional of respiratory epithelium — The working's investigators hypothesis is that the morphology and functional of the epithelium of children with ADV or RV respiratory infection is different between those who progress to PIBO and those who do not.

SUMMARY:
Bronchiolitis obliterans (BO) is an irreversible chronic obstructive pulmonary pathology leading to obstruction and/or obliteration of the small airways. In children, the most common form of BO occurs following a serious lower respiratory tract infection. This is a rare complication; the incidence is unknown. The diagnosis, often late, is made on clinical, spirometric and radiological arguments. The pathophysiology would be linked to damage to the airway epithelium. PIBO is most commonly associated with adenovirus (ADV) infection (serotypes 3, 7, 11 and 21) but also other viruses such as rhinovirus (RV). The treatment of PIBO is not clearly established, it remains empirical.

The research hypothesis is that the morphology of the nasal epithelium of children with ADV or RV infection is different for those progressing to PIBO. The main objective of the proposed observational study is to characterize damage to the respiratory epithelium in these children.

This is a single-center prospective longitudinal study (AP-HM), in children aged 1 month to 6 years, comparing children hospitalized for lower respiratory infection by ADV or RV progressing or not to PIBO. All children included will have a nasal swab and brushing on D0. Children developing PIBO will have nasal brushing with bronchial endoscopy with bronchial biopsies and bronchoalveolar washing at the time of PIBO diagnosis and again at M6 in case of partial response to treatment.

This is therefore a pilot study aimed at defining damage to the respiratory epithelium in children with PIBO following an ADV or RV infection and the role of respiratory epithelial cells in PIBO.

ELIGIBILITY:
Inclusion Criteria:

1. Children from 1 month to 6 years hospitalized at the Timone Enfant University Hospital
2. Diagnosis of an adenovirus or rhinovirus respiratory infection confirmed on a nasal swab, made upon arrival as part of the child's initial care
3. Consent form read, understood, approved and signed by parents before any study procedure
4. Affiliation to a social security scheme or beneficiary of such a scheme

The inclusion criteria for children who were not hospitalized when diagnosed with an adenovirus and rhinovirus respiratory infection at the Timone Enfant University Hospital are:

1. Children from 1 month to 6 years old transferred to the Timone Enfant University Hospital
2. Show the following signs:

   has. Clinical: clinical signs persist 6 weeks after a viral infection: tachypnea, wheezing and/or persistent hypoxemia b. Scan: mosaic appearance +/- bronchiectasis, atelectasis vs. +/- EFR if performed: obstructive ventilatory disorder not or only slightly reversible after bronchodilators
3. Consent form read, understood, approved and signed by parents before any study procedure
4. Affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

1. Refusal of participation in the study by the family will be a reason for non-inclusion, as well as in the absence of parental authority.
2. The existence of an underlying chronic pulmonary pathology (e.g. cystic fibrosis, ciliary dyskinesia).
3. A coagulation pathology.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The main objective is to define damage to the respiratory epithelium in children with PIBO following an Adenovirus (ADV) or Rhinovirus (RV) infection. | through study completion, an average of 3 year
  The morphology of the nasal and bronchial epithelia of PIBO will be analysed during the course of the disease both ex vivo and in vitro. Several criteria will be analysed, such as cell composition, thickness and epithelial cohesion during the culture of reconstituted nasal and/or bronchial epithelium, using microscopy.

SECONDARY OUTCOMES:
Looking for pro-inflammatory and antiviral mediators involved in remodelling and epithelial-mesenchymal transition or that may be involved in the development of a PIBO. | through study completion, an average of 3 year
  Dosage pro-inflammatory and antiviral mediators involved in remodeling and epithelial-mesenchymal transition. Level of expression of adenovirus and rhinovirus receptor: CAR, CD46, ICAM-1.
Evaluating the response of the nasal epithelium to viral stimulation in children with and without PIBO and those who had not developed PIBO after respiratory infection with ADV and/or RV. | through study completion, an average of 3 year
  Quantifying the production of pro-inflammatory mediators with alarmins (TSLP, IL-33 and IL-25), cytokines (IL-6 and IL-8) and antivirals (IFN types I and III).
  TSLP, IL-33, IL-25, IL-6 and IL-8, IFN types I and III will have the same units of measure.
  Assay of PANoptosis markers with apoptosis, pyroptosis and necroptosis: caspase, GSDMD, MKL.
Describing the transcriptomic profile of bronchial biopsies from children with PIBO. | through study completion, an average of 3 year
  An analysis of the transcriptome at the single-cell level will highlight the cellular heterogeneity of bronchial biopsies from children with OPDP, identify rare cell sub-populations and monitor the dynamics of cell evolution during development or as a function of its environment (cell interactions, pathogens, treatments, etc) by comparing them with databases of 'control' biopsies (FasteQ, Hu-man cell lungatlas).
Following the morphology of the nasal and bronchial epithelia of PIBO over the course of the disease | through study completion, an average of 3 year
  Quantifying the production of pro-inflammatory mediators matory with alarmins (TSLP, IL-33 and IL-25), IL-6 and IL-8) and antivirals (IFN types I and III) with ELISA and western blot, involved in remodeling and epithelial-mesenchymal transition (FGF, EGF, TGF-alpha).

CONTACTS AND LOCATIONS:
Overall Officials: Julie MAZENQ, PhD, Principal Investigator — APHP Marseille
Locations (1):
- APHM, Marseille, France